CLINICAL TRIAL: NCT06635083
Title: Comparison of the Effects of Vacuum Bell Therapy and Additional Telerehabilitation on Physical Fitness, Respiratory Functions, Posture and Psychosocial Factors in Children with Pectus Excavatum : a Single-Blind Randomized Controlled Trial
Brief Title: Investigation of the Effectiveness of Telerehabilitation Training in Pectus Excavatum Deformity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMU-FTR-BA-01
Record Dates: First submitted 2024-08-26; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Pectus Excavatum
Keywords: Telerehabilitation; Posture; Congenital Abnormalities; Quality of Life; Physical Fitness; Respiratory Function Tests
MeSH Terms: conditions — Funnel Chest; Congenital Abnormalities | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: Quasi-experimental single-blind randomized comparative study
Who Masked: Outcomes Assessor
Masking Description: Participants with pectus excavatum deformity between the ages of 10 and 14 who apply to the clinic where the study will be conducted by dividing into two groups using the random allocation software computer program.The outcomes assessor will not know which groups individuals assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vacuum bell therapy (Active Comparator): This group will use a vacuum bell for one hour in the morning and evening, as recommended by an experienced thoracic surgeon.
  Interventions: Other: Telerehabilitation
- Vacuum bell therapy+telerehabilitation (Experimental): Telerehabilitation based exercises and vacuum bell therapy will be applied to this group. Video conference software system will be installed on the subjects' laptops or tablets. After the evaluations, exercises will be taught to the individuals in the clinic. Then, the following exercises will be done with the physiotherapist via video conference 3 sessions per week.
  Interventions: Other: Telerehabilitation

INTERVENTIONS:
Other: Telerehabilitation — A video conference software system will be installed on the subjects' laptops or tablets. Then, via video conference, strengthening/stretching exercises and breathing exercises will be performed for the areas affected by the deformity with the physiotherapist three times a week.

SUMMARY:
The aim of this study is to investigate the effectiveness of telerehabilitation-based exercise training in addition to Vacuum Bell therapy on physical fitness, respiratory functions, posture and psychosocial factors in boys aged between 10-14 years diagnosed with pectus excavatum.

DETAILED DESCRIPTION:
Pectus excavatum (PE) is the most common congenital chest wall deformity. It is seen in approximately 1 in 400 live births. PE is characterized by varying degrees of depression of the sternum and rib cartilage. Although its etiopathogenesis is not fully understood, it is thought to be caused by intrauterine pressure on the sternum from an abnormal fetal position, sequelae of diseases such as syphilis and rickets, muscle imbalances in the anterior diaphragm that pull the xiphoid and sternum backwards, and abnormal growth of the costal cartilage junction between the rib and the sternum.

In a typical PE, the lower 1/3 of the sternum and adjacent costal cartilages are seen to collapse. Children with PE are usually tall and have abnormal posture. Scoliosis has been diagnosed in approximately 29% of children with PE. Studies have shown that the most common posture disorders in children with PE are; head forward posture, rounded shoulders, thoracic kyphosis, winged scapula and anterior rotation of the pelvis. In children with PE; decreased flexibility of the upper trapezius, scalene, sternocleidomastoid, pectoralis major muscles; loss of strength in the back extensors, abdominals, quadratus lumborum, lower/middle part of the trapezius and rhomboids have been reported. In addition to orthopedic problems; psychosocial problems related to physical appearance such as body image anxiety, social isolation, introversion, shyness, anxiety and depression have also been detected. It has been predicted that restriction of activities, poor posture and avoidance of sports activities due to deterioration of physical appearance may lead to weakness and other problems in the musculoskeletal system. In addition, it has been published that the cardiovascular endurance of adolescents with moderate and severe PE is lower than that of healthy controls, causing these patients to have reduced physical activity. In recent years, conservative treatment approaches have been increasing. The main conservative treatment methods applied for these patients are vacuum bell treatment, orthosis and physiotherapy. A rehabilitation program planned according to the needs of the person can help increase the quality of life of the individual with PE. Studies have reported that various exercise applications contribute to a decrease in deformity and positive developments in posture. Telerehabilitation is defined as a rehabilitation method carried out remotely between the patient and the health professional through telecommunication technologies such as telephone, internet, and video conference. Telerehabilitation methods can be quite effective in terms of high participation and compliance rates, behavioral changes in lifestyle, the opportunity for the patient to receive rehabilitation in their own environment, the chance to benefit from rehabilitation for a longer period of time and cost efficiency. In addition, the rate at which the rehabilitation program is affected by the low number of specialists in the geography where the patient lives, the lack of transportation facilities and physical disabilities is minimized thanks to telerehabilitation. Accessibility, flexible hours that can adapt to children's busy school programs and time savings, the opportunity for the participation of their families and the interest of children in technology are thought to motivate them to participate in treatment. In the literature study, no study was found showing the effectiveness of exercise training applied with telerehabilitation in children with pectus excavatum deformity. The purpose of this study is to examine the effectiveness of telerehabilitation-based exercise training applied in addition to Vacuum Bell treatment on physical fitness, respiratory functions, posture and psychosocial factors in boys between the ages of 10-14 diagnosed with pectus excavatum.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 10-14
* Boys
* Those who have undergone Vacuum Bell treatment for the first time

Exclusion Criteria:

* Those with complex type pectus deformity
* Those who have undergone any surgical treatment due to pectus excavatum
* Those with chronic systemic disease (cardiovascular, gastrointestinal, metabolic)
* Those with diagnosed serious psychiatric disease
* Those with scoliosis over 20 degrees
* Those with other musculoskeletal anomalies and connective tissue disorders (Marfan syndrome, Turner syndrome, neurofibromatosis tuberous sclerosis)
* Those with neurological disease
* Those with hearing or vision impairment that cannot be corrected with hearing aids or glasses
* Those who do not have internet access or do not own a tablet/computer

Ages: 10 Years to 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Estimated)
Dates: Start 2024-10-10 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Physical Fitness | 6 months
  Health-Related Physical Fitness
  Health-related physical fitness will be assessed using the FITNESSGRAM® test battery. This test battery was developed to record the abilities of his children.
  Health-related physical fitness components:
  * Aerobic capacity
  * Body composition
  * Strength
  * Endurance
  * Flexibility

SECONDARY OUTCOMES:
Pulmonary functions | 6 months
  Pulmonary functions will be assessed by two devices.
  1. Forced Expiratory Volume in 1 Second (FEV1) Forced Vital Capacity (FVC) Voluntary Ventilation (MVV) will be measured by a portable spirometer device.
  2. Peak Expiratory Flow (PEF) will be measured by Peak Flow Meter

OTHER OUTCOMES:
Posture | 6 months
  Posture assessment will be done by lateral photography. Photographs will be taken from 90 degrees sideways and 1.5 meters away with a digital camera placed on a tripod. Markers will be placed on certain anatomical points (eye canthus, ear tragus, acromion, spinous process of the 7th cervical vertebra, spinous processes of the 4th and 7th thoracic vertebrae, spinous process of the 1st lumbar vertebra, spina iliaca anterior superior (SIAS), trochanter major, lateral of the midpoint of the knee joint) and angular calculations will be made from the lateral projection of these points.
Handgrip strength | 6 months
  It has been reported that it is strengthened with general body muscle strength. Therefore, it is widely used because it is a cheap, practical and easy method for determining general body muscle strength. During this test, subjects will be asked to make a baseline in sitting positions, with the elbow in 90 degree flexion, the shoulder in adduction and the forearm in neutral position. For this reason, the average and value repeated three times will be recorded.
Body Image Perception | 6 months
  Body Image Assessment
  This scale aims to measure the individual&amp;amp;amp;amp;amp;amp;#39;s level of satisfaction of their body. This scale includes a total of 40 items with scores between 1 and 5. A higher score indicates a higher level of body image satisfaction.
Social Anxiety | 6 months
  Social Anxiety Scale for Children
  Social anxiety will be assessed using the 'Social Anxiety Scale for Children-Revised, a self-report designed to assess social fears in children. The items selected in anxiety scales developed for children are related to social situations.
Psychological State | 6 months
  This assessment will be made using the 'Depression Scale for Children. 27-question scale and each item is scored between 0-2. A high total score indicates a high level of depression. The pathology cut-off point was determined as 19 points.
Quality of life assessment | 6 months
  Quality of Life Assessment The Turkish version of the Nuss Questionnaire, a disease-specific health-related quality of life assessment tool for patients with pectus deformities, will be used to assess the quality of life of patients and their parents. The total scores of patients on the form range from 12 to 48, while the total scores of parents&amp;amp;amp;amp;#39; forms range from 11 to 44. Higher scores indicate better overall satisfaction and better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Emine H Tüzün, Study Director — Eastern Mediterrenian University
Locations (1):
- Marmara Üniversitesi Pendik Eğitim Ve Araştirma Hastanesi, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No